CLINICAL TRIAL: NCT03627338
Title: Medikamentenadhärenz Bei Patientinnen Und Patienten Mit Leberzirrhose
Brief Title: Medication Adherence in Patients With Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: HannoverGAS-Adhaerenzprojekt
Record Dates: First submitted 2018-07-26; First posted 2018-08-13 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Norfloxacin: evaluate medication adherence, patient history, medication beliefs and medication satisfaction, depression, anxiety and health-related quality of life
  Interventions: Diagnostic Test: questionaire, interview
- Non-selective beta blockers: evaluate medication adherence, patient history, medication beliefs and medication satisfaction, depression, anxiety and health-related quality of life
  Interventions: Diagnostic Test: questionaire, interview
- diuretics: evaluate medication adherence, patient history, medication beliefs and medication satisfaction, depression, anxiety and health-related quality of life
  Interventions: Diagnostic Test: questionaire, interview

INTERVENTIONS:
Diagnostic Test: questionaire, interview — questionaire, interview

SUMMARY:
With this unfunded, investigator-initiated prospective, observational, explorative, single-arm and diagnostic single-centre study the investigators aim to evaluate medication adherence in patients with advanced liver cirrhosis

DETAILED DESCRIPTION:
The main objective of the study is to investigate drug adherence in cirrhotic patients and to gain a better understanding of the causes of deficient adherence including evaluation for medication beliefs, satisfaction, depression, anxiety and health-related quality of life. A number of long-term medications have been approved for this group of patients in various indications and / or recommended by guidelines. However, adherence has not been adequately investigated yet. The investigators aim to focus on the following groups of ingredients / classes:

* Primary and secondary antibiotic prophylaxis (e.g. Norfloxacin)
* Non-selective beta-blockers (e.g. Carvedilol and Propranolol)
* diuretics (Spirolactones [e.g. Spironolacton], loop diuretics) Methodically, this is will be investigated in particular by taking into account the patients history, standardized questionnaires and validated interviews.

ELIGIBILITY:
Inclusion Criteria:

* Treatment at Dept. of Gastroenterology, Hepatology and Endocrinology at Med. School of Hannover
* Liver cirrhosis
* Written consent for the use of personal data and health data for the purpose of this study

Exclusion Criteria:

* lack of written consent
* No consent ability
* Lack of literacy
* Inadequate knowledge of German language

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In addition to inclusion criteria: Treatment with Norfloxacin, Non-selective beta blockers and/or diuretics
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Medication adherence with BAASIS | One-point first visit, cross-section-designed study during the 24 month study period
  Medication adherence will be investigated by using the BAASIS interview ((Basel Assessment of Adherence with Immunosuppressive Medication Scale)) The investigators use a validated German version of this instruments. Adherence is classified by means of a reliable rating system. For the BAASIS: Any YES on any of the questions 1a, 1B, 2 or 3 indicates an issue with implementation."YES" on item 4 indicates non-persistence of medication use. For the BAASIS the Overall can be quantified with both ways: as a dichtomus variable or as a continuous variable. The dichotomous variable of the BAASIS will use the scores on the questions assessing implementation and persistence (Questions 1a, 1b, 2, 3 and 4). The continuous variable will use a Visual Analogue Scale (VAS) assessing overall medication adherence over the last 4 weeks with higher scores represent higher perceived overall adherence.
Medication adherence with MARS | One-point first visit, cross-section-designed study during the 24 month study period
  Medication adherence will be investigated by using the MARS ("Medication Adherence Report Scale" ) questionnaire (self-report). The investigators use a validated German version of this instruments. Adherence is classified by means of a reliable rating system. This 5-items scale asks respondents to rate the frequency with which they engage in each of 5 aspects of non-adherent behaviour Eg deciding to miss a dose, forgetting to take a dose), rated on a five point scale (where 5=never, 4 = rarely, 3 = sometimes, 2 = often and 1= very often). Scores for each of the 5 items were summed to give a scale score ranging from 5 to 25, where higher scores indicate higher levels of reported adherence.
  Adherence can be expressed as a continuous scale, or by separating into 'high' and 'low' adherence groups on the basis of scale scores.

SECONDARY OUTCOMES:
Medication satisfaction | One-point first visit, cross-section-designed study during the 24 month study period
  Medication satisfactions is evaluated by using a self-report validated 19-item questionnaire ; the SIMS-D ("Satisfaction with Information about Medicines Scale"). Mediaction satisfaction is classified by means of a reliable rating system.
Medication belief | One-point first visit, cross-section-designed study during the 24 month study period
  The investigators will use the "Beliefs about Medicines Questionnaire" (BMQ) as reliable survey tool for recording drug-related beliefs and perceptions of their benefits and / or harms. For this projects the investigators will use most recent German version authored by Nestoriuc et al. The BMQ is divided into a general and a drug-specific section. Medication belief is classified by means of a reliable rating system.
Depression | One-point first visit, cross-section-designed study during the 24 month study period
  Depression will be evaluated by another self-reported instrument, the "Patient Health Questionnaire" (PHQ 9), which is a screening tool for depression disorders with a sufficient reliability. Depression is classified by means of a reliable rating system.
Anxiety | One-point first visit, cross-section-designed study during the 24 month study period
  The investigators will use GAD 7 ("Generalized Anxiety Disorder Screeners"), another questionnaire, to screen for general anxiety disorders. This refers to the last 2 weeks and covers the most important clinical criteria according to DSM-IV. Anxiety is classified by means of a reliable rating system.
health-related Quality of Life | One-point first visit, cross-section-designed study during the 24 month study period
  In addition, the investigators will use the CLDQ "Chronic Liver Disease Questionnaire" to examine the health-related quality of life in patients with hepatopathy regardless of severity or aetiology with high reliability. HRQoL is classified by means of a reliable rating system. The scale values of the subject are obtained by assigning 1 (always), 2 (mostly), 3 (common), 4 (repeated), 5 (sometimes), 6 (rare) and 7 (never)points. The values of the subscales of the original version are obtained by adding the items of the respective scale on the CLDQ-D evaluation sheet. The range of possible values per scale is between 1 and 7. Normative values of a representative population sample are not available. For comparison, the results of clinical trials can be used. Low values mean a reduced, high values a good health-related quality of life
Medication knowledge | One-point first visit, cross-section-designed study during the 24 month study period
  At last, the investigators will evaluate the participant knowledge about their medication by using a self-constructed questionnaire. For this purpose we constructed an own Rating System.
Sociodemographic data | One-point first visit, cross-section-designed study during the 24 month study period
  Sociodemographic data (e.g. age, education, income) will be collected with another self-constructed questionnaire in addition to already collected data of patients history from the disease record

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Maasoumy, Associate Professor, MD, Principal Investigator — Medical School of Hannover
Locations (1):
- Medical School of Hannover, Hanover, Germany

IPD SHARING:
Plan to Share IPD: Undecided